CLINICAL TRIAL: NCT04006236
Title: Growth and Tolerance of Infants Fed Extensively Hydrolyzed Casein-Based Infant Formulas
Brief Title: Infants Fed Extensively Hydrolyzed Casein-Based Infant Formulas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AL33
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Infant Development

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Infant Formula (Experimental): extensively hydrolyzed casein protein
  Interventions: Other: Experimental Infant Formula
- Control Infant Formula (Active Comparator): extensively hydrolyzed casein protein
  Interventions: Other: Control Infant Formula

INTERVENTIONS:
Other: Experimental Infant Formula — Feed Ad Libitum
  Arms: Experimental Infant Formula
Other: Control Infant Formula — Feed Ad Libitum
  Arms: Control Infant Formula

SUMMARY:
This is a randomized, controlled, double-blind, multicenter parallel study to evaluate the growth, tolerance and compliance of healthy infants fed infant formulas with extensively hydrolyzed casein protein.

ELIGIBILITY:
Inclusion Criteria:

* Participant is judged to be in good health
* Participant is a singleton from a full-term birth with a gestational age of 37-42 weeks
* Participant's birth weight was > 2490 g (~5 lbs. 8 oz.)
* Parent(s) confirm their intention to feed their infant the study product as the sole source of nutrition for the duration of the study
* Parent(s) confirm their intention not to administer vitamins, minerals (with the exception of Vitamin D supplements), solid foods or juices to their infant from enrollment throughout the duration of the study
* Participant's parent(s) has voluntarily signed and dated an Informed Consent Form (ICF), approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) and provided Health Insurance Portability and Accountability Act (HIPAA) (or other applicable privacy regulation) authorization

Exclusion Criteria:

* An adverse maternal, fetal or participant medical history that is thought by the investigator to have potential for effects on tolerance, growth, and/or development.
* Participant is taking and plans to continue taking medications, home remedies, prebiotics, probiotics, herbal preparations or rehydration fluids that might affect gastrointestinal (GI) tolerance
* Participant participates in another study that has not been approved as a concomitant study by AN.
* Participant has an allergy or intolerance to any ingredient in the study product
* Participant has been treated with antibiotics within 1 week prior to enrollment

Ages: 0 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 245 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Weight | Day of Age (DOA) 14 to 119
  Interval weight gain per day

SECONDARY OUTCOMES:
Length | Study Day (SD) 1 to DOA 119
  Interval length gain per day
Head Circumference | Study Day (SD) 1 to DOA 119
  Interval HC gain per day
Stool Characteristics | Study Day (SD) 1 to DOA 119
  Parent Completed Diary
Formula Intake | Study Day (SD) 1 to DOA 119
  Parent Completed Diary

OTHER OUTCOMES:
Infant Feeding and Stool Patterns Questionnaire | Exit or DOA 119
  Parent completed questionnaire; 16 questions with 5 categories scaled in the negative direction
Infant Behavior Questionnaire | Exit or DOA 119
  Parent completed questionnaire; 22 questions with 5 categories scaled in the negative direction
Formula Satisfaction Questionnaire | Exit or DOA 119
  Parent completed questionnaire; 13 questions of up to 5 categories scaled in the negative direction

CONTACTS AND LOCATIONS:
Overall Officials: Carlett Ramirez, Study Chair — Abbott Nutrition
Locations (17):
- United States (17):
  - MedPharmics, LLC, Phoenix, Arizona
  - Watching Over Mothers & Babies, Tucson, Arizona
  - Paramount Research Solutions, College Park, Georgia
  - Springs Medical Research, Owensboro, Kentucky
  - MedPharmics, LLC, Metairie, Louisiana
  - MedPharmics, LLC, Gulfport, Mississippi
  - Quality Clinical Research Inc, Omaha, Nebraska
  - MedPharmics, LLC, Albuquerque, New Mexico
  - PMG Research of Peidmont Healthcare, Statesville, North Carolina
  - Pediatric Associates of Fairfield, Inc., Fairfield, Ohio
  - Institute of Clinical Research, LLC, Mentor, Ohio
  - The Cleveland Pediatric Research Center, LLC, Middleburg Heights, Ohio
  - Children's Hospital, Sioux Falls, South Dakota
  - Midsouth Center for Clinical Research, Memphis, Tennessee
  - Ventavia Research Group, Llc, Fort Worth, Texas
  - Ventavia Research Group, Houston, Texas
  - Ventavia Research Group, LLC, Plano, Texas

IPD SHARING:
Plan to Share IPD: No